CLINICAL TRIAL: NCT06887868
Title: Immediate Effect of Mobilization with Movement on Squat Self-reported Functional Ability, Pain Intensity, and Pain-free Range of Motion in People with Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Immediate Effect of Mobilization with Movement on Squat Self-reported Functional Ability, Pain Intensity, and Pain-free Range of Motion in People with Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Daniela Ferreira Carneiro, MSc, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE2023/17
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Knee Osteoarthritis; manual therapy; mobilization with movement; functional status; Mulligan concept; neurophysiological effect
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MWM (Experimental): The intervention group received the MWM technique, which involved the manual application of a sustained translational or rotational glide force, either medial or lateral, on the tibia, while an active partial weight-bearing lunge movement was performed. All glide forces were tested in a randomly pre-established order, and the most effective force for symptom relief and improvement in knee range of motion was selected for the intervention.
  Interventions: Procedure: Mobilization with movement
- Sham MWM (Sham Comparator): In the sham group, the participants underwent a similar procedure to those in the intervention group. The physiotherapist mimicked the pain-reducing glide direction without applying glide force while the participants performed the active lunge movement. To achieve this, the physiotherapist's hands lightly touched the knee skin, with one hand on the tibia and the other on the femur over the joint surfaces. The volume of the sham MWM technique was identical to that of the MWM technique administered to the intervention group.
  Interventions: Procedure: Sham mobilization with movement

INTERVENTIONS:
Procedure: Mobilization with movement — Manual application of a sustained translational or rotational glide force, either medial or lateral, on the tibia, while an active partial weight-bearing lunge movement was performed.
  Other Names: MWM; Mulligan concept
  Arms: MWM
Procedure: Sham mobilization with movement — The physiotherapist mimicked the pain-reducing glide direction without applying glide force while the participants performed the active lunge movement. To achieve this, the physiotherapist's hands lightly touched the knee skin, with one hand on the tibia and the other on the femur over the joint surfaces.
  Arms: Sham MWM

SUMMARY:
Mobilization with movement (MWM) appears to reduce pain, improve knee range of motion, and enhance physical functioning in individuals with knee osteoarthritis (KOA). However, it remains unclear whether the severity grading of structural damage in KOA affects its effects. This study aims to analyze the immediate effect of MWM on squat self-reported functional ability, pain intensity, and pain-free range of motion in people with KOA, and to verify it its effect is influenced by the severity grading of structural damage.

ELIGIBILITY:
Inclusion Criteria:

* male or female;
* aged over 45 years;
* clinically diagnosed with symptomatic unilateral KOA, classified as grade 1-3 according to the Kellgren and Lawrence system;
* fulfilled the classification criteria of the American College of Rheumatology for KOA;
* reported frequent episodes of pain in the knee joint during sit-to-stand movements for at least 3 months.

Exclusion Criteria:

* had KOA secondary to rheumatoid arthritis and other inflammatory and autoimmune conditions;
* reported lumbar pain radiating to the knee or lumbar pain as the primary complaint;
* had a history of knee or lower limb surgery;
* had a systemic or local infection;
* had received an intra-articular corticosteroid or hyaluronic acid injection within the past 6 months;
* reported current or past (within 4 weeks) oral corticosteroid use;
* had any condition in the lower limbs that would prevent performing the deep squat test;
* had clinical conditions in which manual therapy is generally contraindicated (such as fracture, osteoporosis, instability, infectious arthritis, tumors, joint ankylosis, acute inflammatory disorders, or lack of a diagnosed joint lesion).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Functional ability | Baseline
  The Patient-Specific Functional Scale was used to assess self-reported functional ability. This scale is a self-reported, valid, and responsive outcome measure used to quantify activity limitations and evaluate functional outcomes for individuals with musculoskeletal conditions. Participants rated their current level of ability to performing the deep squat test on an 11-point scale at a level experienced prior to injury or change in functional status, where "0" represents "unable to perform" and "10" represents "able to perform at prior level.
Knee Pain | Baseline
  The Numeric Pain Rating Scale is a self-reported, valid, and responsive outcome measure that was used in this study to quantify pain intensity. Participants rated their current pain intensity related to performing the deep squat test on a scale divided into eleven equal parts, numbered consecutively from 0 to 10, where "0" represents "No Pain" and "10" represents "Worst Possible Pain" (the most intense pain imaginable).
Pain free Range of Motion (ROM) | Baseline
  This test has been advocated as a useful method for evaluating knee pain and function. Participants began the deep squat test by standing with their feet flat on the floor, approximately shoulder-width apart, aligned in the sagittal plane, and their hands placed on their pelvis (adapted from the original test description). They were then instructed to squat (buttocks towards the heels) as low as possible until the onset of pain, while maintaining an upright torso, avoiding asymmetric weight shift, and keeping their heels and toes in position. Before the test, participants viewed a demonstration video to optimize their understanding of the procedures. Additionally, they were given the opportunity to perform a practice trial of the deep squat test at a pain-free range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- E2S | P.PORTO - Escola Superior de Saúde do Politécnico do Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No